CLINICAL TRIAL: NCT00326625
Title: A Multinational, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Assess the Efficacy, Tolerability and Safety of 40 mg Glatiramer Acetate Injection in Subjects With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Clinical Trial of Glatiramer Acetate in Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Pharmaceutical Industries, Ltd. (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALS-GA-201
Record Dates: First submitted 2006-05-16; First posted 2006-05-17 (Estimated); Results first posted 2021-10-20 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Glatiramer Acetate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 40 mg glatiramer acetate (GA) (Experimental): Pre-filled syringe of 40 mg glatiramer acetate (GA) for injection, administered subcutaneously once a day.
  Interventions: Drug: 40 mg glatiramer acetate
- Placebo (Placebo Comparator): Pre-filled syringe of matching placebo, administered subcutaneously once a day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 40 mg glatiramer acetate — parenteral drug
  Arms: 40 mg glatiramer acetate (GA)
Drug: Placebo
  Arms: Placebo

SUMMARY:
Teva is developing 40 mg/ml Glatiramer Acetate (GA) Injection , administered once daily under the skin, for the treatment of ALS. The study drug is a higher dose formulation of Copaxone® (20 mg/ml GA), a marketed medication, approved for the treatment of relapsing-remitting multiple sclerosis. GA is an immunomodulating drug that has anti inflammatory and neuroprotective properties, which are believed to be of therapeutic value in ALS. The study treatment duration is 1 year (52 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of definite or probable ALS in accordance with the El-Escorial criteria.
2. Subject has experienced his/her first ALS symptoms within 3 years prior to the screening visit.
3. Slow VC test equal or greater than 70% of the predicted value.
4. The sum of the 3 respiratory items on the ALSFRS-R must total at least 10 points.
5. Stable dose of riluzole for at least 8 weeks prior to screening.
6. Age - 18-70 (inclusive).

Exclusion Criteria:

1. The use of invasive or non-invasive ventilation.
2. Subject having undergone gastrostomy.
3. Subject with any clinically significant or unstable medical condition.
4. Subjects participating in any other clinical trial (within 12 weeks prior to screening and thereafter).
5. Additional criteria per protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2006-07-27 (Actual); Primary Completion 2008-06-17 (Actual); Study Completion 2008-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merav Bassan, PhD., Study Chair — Teva Pharmaceuticals Industries LTD
Locations (7):
- Belgium (2):
  - Teva Benelux, Haarlem
  - Teva Benelux, Leuven
- Teva France, Paris, France
- Teva Germany, Mörfelden-Walldorf, Germany
- Teva Israel, Tel Aviv, Israel
- Teva Italy, Milan, Italy
- Teva UK, Aylesbury, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 366 participants were randomized in a 1:1 ratio to one of two treatment groups, Glatiramer Acetate 40 mg or matching placebo. The study duration was 52 weeks with a follow up period of up to 44 weeks.
Groups:
- Glatiramer Acetate 40mg: Pre-filled syringe of 40 mg glatiramer acetate (GA) for injection, administered subcutaneously once a day
Period: Overall Study
Arm/Group | Glatiramer Acetate 40mg | Placebo
Started | 184 | 182
Completed | 130 | 144
Not Completed | 54 | 38
Not completed — Adverse Event | 20 | 9
Not completed — Withdrawal by Subject | 15 | 12
Not completed — Death | 18 | 16
Not completed — Lost to Follow-up | 1 | 0
Not completed — prescheduled medical intervention | 0 | 1

BASELINE CHARACTERISTICS:
Population: The intent to treat (ITT) analysis set included all randomized participants who took at least one dose of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Glatiramer Acetate 40mg | Placebo | Total
Number analyzed (Participants) | 184 | 182 | 366
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.7 (9.6) | 54.7 (9.6) | 55.2 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 72 | 141
  Male | 115 | 110 | 225
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 182 | 182 | 364
  Black or African American | 1 | 0 | 1
  Hispanic | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Slope of Change From Baseline in the ALS Functional Rating Scale (ALSFRS-R)
Description: The ALSFRS-R is a questionnaire-based scale for monitoring the progression of disability in patients with ALS. It is composed of 12 items, each scored between 0 and 4.The total score, calculated as the sum of these 12 items, ranges from 0 to 48. The higher the score, the less disabled the participant. Timepoints after baseline were included in calculation of slope of change in ALSFRS-R. Slope is derived from the time by treatment interaction term from the Repeated Measures Analysis of Covariance model. Descriptive statistics of the slope are reported.
Time Frame: Baseline, Weeks 4, 8, 12, 17, 22, 26, 31, 36, 40, 44, 48, 52
Population: The intent-to-treat (ITT) analysis set consisted of all randomized participants who took at least one dose of the study drug.
Measure: Mean (Standard Error); unit: Units on a Scale per Month
Arm/Group | Glatiramer Acetate 40mg | Placebo
Number analyzed (Participants) | 184 | 182
Units on a Scale per Month | -1.05 (0.059) | -1.00 (0.058)
Statistical Analysis 1: Comparison: Glatiramer Acetate 40mg vs Placebo; Analysis compares the ALSFRS-R slopes of change from baseline between treatment groups. Analysis includes the following covariates: time from randomization, treatment group, time by treatment interaction, center, Riluzole use, age, site of ALS onset, time from ALS onset and baseline ALSFRS-R score; Test type: Superiority; p = 0.4807, ANCOVA; Slope difference = -0.06, 95% CI 2-sided [-0.22 to 0.10], Standard Error of Mean 0.083 — Glatiramer acetate vs. Placebo

2. Secondary Outcome: Time to Event: Death, Tracheostomy, Permanent Assisted Ventilation
Description: Composite endpoint of time to death, tracheostomy, or permanent assisted ventilation analyzed using the Cox's proportional hazards model to compare the risk of death, tracheostomy, or permanent assisted ventilation between treatment groups. The model includes center country, Riluzole© use, site of ALS onset, time from ALS onset, and baseline ALSFRS-R score, baseline slow VC and baseline BMI as covariates. Because less than 50% of participants experienced the event, the median time to event (i.e. the descriptive statistic for the day for which 50% of participants experienced the event) could not be calculated. Hence the days are reported as not available.
Time Frame: Baseline up to 52 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Glatiramer Acetate 40mg | Placebo
Number analyzed (Participants) | 184 | 182
Days | NA [NA to NA] — Median days to event could not be calculated because less than 50% of participants experienced the event. Hence the days are reported as NA. | NA [NA to NA] — Median days to event could not be calculated because less than 50% of participants experienced the event. Hence the days are reported as NA.
Statistical Analysis 1: Comparison: Glatiramer Acetate 40mg vs Placebo; Analysis covariates are center, riluzole use, site of ALS onset, time from ALS onset, baseline ALSFRS-R score, baseline slow vital capacity (VC) and baseline body mass index (BMI); Test type: Superiority; p = 0.8583, Regression, Cox; Hazard Ratio (HR) = 1.060, 95% CI 2-sided [0.560 to 2.005] — Glatiramer acetate vs. Placebo

ADVERSE EVENTS:
Time Frame: Baseline up to 96 weeks.
Description: The safety analysis set included all participants that took at least one dose of study drug.
Arm/Group | Glatiramer Acetate 40mg | Placebo
All-Cause Mortality (participants affected / at risk) | 22/184 | 17/182
Serious Adverse Events (participants affected / at risk) | 55/184 | 54/182
Other Adverse Events (participants affected / at risk) | 167/184 | 133/182
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glatiramer Acetate 40mg (N=184) | Placebo (N=182)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 2 (2) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cyanosis (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 6 (6) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Catheter site haemorrhage (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 2 (2)
Chills (General disorders) | 1 (1) | 0 (0)
Condition aggravated (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 1 (1)
Disease progression (General disorders) | 1 (1) | 0 (0)
General physical health deteriora (General disorders) | 0 (0) | 1 (1)
Hyperthermia (General disorders) | 2 (2) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Type IV hypersensitivity reaction (Immune system disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 2 (3) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (2)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 7 (8) | 7 (7)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (3)
Bone fissure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 4 (5) | 4 (6)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pneumocephalus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increas (Investigations) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1)
Coma (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (2) | 1 (1)
Meningorrhagia (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary dis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 7 (8)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 4 (5)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Increased viscosity of bronchial (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 15 (16) | 18 (21)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Endotracheal intubation (Surgical and medical procedures) | 0 (0) | 1 (1)
Gastrostomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Haemorrhoid operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Laparotomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Laryngeal polypectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Mechanical ventilation (Surgical and medical procedures) | 0 (0) | 2 (2)
Tracheostomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 2 (2) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glatiramer Acetate 40mg (N=184) | Placebo (N=182)
Constipation (Gastrointestinal disorders) | 18 (18) | 14 (15)
Diarrhoea (Gastrointestinal disorders) | 17 (23) | 13 (18)
Dysphagia (Gastrointestinal disorders) | 11 (12) | 9 (10)
Nausea (Gastrointestinal disorders) | 17 (20) | 11 (12)
Fatigue (General disorders) | 11 (11) | 14 (15)
Injection site erythema (General disorders) | 80 (239) | 9 (11)
Injection site induration (General disorders) | 24 (24) | 1 (1)
Injection site mass (General disorders) | 15 (16) | 0 (0)
Injection site nodule (General disorders) | 11 (58) | 1 (1)
Injection site pain (General disorders) | 52 (81) | 8 (8)
Injection site pruritus (General disorders) | 46 (181) | 3 (3)
Injection site swelling (General disorders) | 24 (72) | 0 (0)
Malaise (General disorders) | 10 (16) | 5 (8)
Oedema peripheral (General disorders) | 5 (5) | 10 (11)
Bronchitis (Infections and infestations) | 12 (14) | 19 (20)
Nasopharyngitis (Infections and infestations) | 31 (38) | 30 (40)
Upper respiratory tract infection (Infections and infestations) | 10 (12) | 9 (12)
Urinary tract infection (Infections and infestations) | 8 (10) | 10 (14)
Fall (Injury, poisoning and procedural complications) | 37 (65) | 45 (105)
Back pain (Musculoskeletal and connective tissue disorders) | 18 (20) | 15 (15)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 (12) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 11 (18) | 18 (26)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 13 (13) | 12 (12)
Dizziness (Nervous system disorders) | 12 (14) | 6 (6)
Headache (Nervous system disorders) | 23 (32) | 27 (33)
Anxiety (Psychiatric disorders) | 10 (11) | 5 (5)
Depression (Psychiatric disorders) | 9 (9) | 16 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 12 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 (26) | 8 (9)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 11 (12)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 11 (15) | 7 (7)
Flushing (Vascular disorders) | 14 (19) | 2 (2)
Hot flush (Vascular disorders) | 16 (27) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.